CLINICAL TRIAL: NCT03245216
Title: Facilitating Motor Skill Learning by Aerobic Training in Parkinson's Disease
Brief Title: Facilitating Motor Skill Learning in Parkinson's Disease
Acronym: FAST-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: German Foundation for Neurology (Other); Department of Molecular Neurology, Faculty of Medicine, University Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Simon Steib, PhD, Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DSN-032017
Record Dates: First submitted 2017-07-31; First posted 2017-08-10 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; motor learning; aerobic exercise; cardiovascular exercise; balance; postural instability; motor skill
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise + motor skill practice (Experimental): acute bout of aerobic exercise before motor learning
  Interventions: Behavioral: aerobic exercise; Behavioral: motor learning
- rest + motor skill practice (Active Comparator): seated rest before motor learning
  Interventions: Behavioral: rest; Behavioral: motor learning

INTERVENTIONS:
Behavioral: aerobic exercise — Single-bout of moderate intensity aerobic exercise on a cycle ergometer before motor learning
  Arms: aerobic exercise + motor skill practice
Behavioral: rest — Seated rest before motor learning
  Arms: rest + motor skill practice
Behavioral: motor learning — Motor learning task on a stability platform (Stabilometer). Participants try to keep the tiltable platform in an horizontal position.

SUMMARY:
The study is designed to assess the effects of aerobic exercise on motor learning in Parkinson patients. Specifically, the investigators examine whether a single bout of moderate intensity aerobic exercise, performed immediately before task practice, facilitates the acquisition and retention of a motor skill. In a cross-over design, participants will be randomly allocated to either the intervention group (aerobic exercise before motor learning) or control group (rest before motor learning).

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disorder that is characterized by motor control impairments, such as gait disturbances and postural instability. Beneficial effects of exercise are attributed to mechanisms of neuroplasticity, and task-specific motor training is consequently considered to be a motor learning process. While motor learning is preserved in persons with Parkinson's disease, slower acquisition rates and reduced retention have been reported compared to healthy individuals.

Thus, it is crucial to identify strategies to enhance motor learning in people with Parkinson's disease. Recent studies have accumulated evidence to show that aerobic exercise can facilitate motor skill learning. However, these observations are limited to healthy individuals and have not been addressed in individuals with neurologic conditions.

The present study is designed to assess the effects of a single bout of moderate intensity aerobic exercise on a motor skill learning task in patients with Parkinson's disease.

In a cross-over design, participants will be randomly allocated to one of two groups. Both groups will practice balancing on a specific stability platform (motor learning task). The experimental group will additionally perform a bout of aerobic exercise (cycle ergometer) immediately before the motor learning task, while the control group will rest before practice. Subsequently, the acquisition and one-day retention of the motor learning task will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 1-3 on Hoehn & Yahr scale
* Ability to stand unaided and walk without an assistive device
* Stable medication during the study period

Exclusion Criteria:

* On-off and wearing-off phenomena
* Unstable medical or psychiatric illness
* Clinically relevant cardiovascular or orthopaedic disease
* Severe polyneuropathy
* Cognitive impairment
* Smoking > 10 cigarettes/day
* Caffeine > 6 cups of coffee/day
* Alcohol > 50 g (two glasses)/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Motor Learning (Precision) | Baseline (first trial of practice day 1), 1 day (last trial of practice day 1), and 7 days (first trial of 7-day retention session).
  Change from baseline in time in balance (±5° from horizontal) during balancing task.

SECONDARY OUTCOMES:
Motor Learning (Variability) | Baseline (first trial of practice day 1), 1 day (last trial of practice day 1), and 7 days (first trial of 7-day retention session).
  Change from baseline in mean standard deviation (root mean square error) of platform deflection (in degree).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Steib, Dr., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Institute of Sport Science and Sport
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Institute of Sport Science and Sport, Gebbertstr. 123b, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steib S, Wanner P, Adler W, Winkler J, Klucken J, Pfeifer K. A Single Bout of Aerobic Exercise Improves Motor Skill Consolidation in Parkinson's Disease. Front Aging Neurosci. 2018 Oct 22;10:328. doi: 10.3389/fnagi.2018.00328. eCollection 2018. PMID 30405397
- See also: project webpage — https://www.sport.fau.de/lehrstuehle-und-fachgebiete/bewegung-und-gesundheit/forschungsprojekte/optimierung-motorischer-lernprozesse-in-der-rehabilitation-von-parkinsonpatienten/